CLINICAL TRIAL: NCT01002963
Title: A Double-Blind (3rd Party Open), Randomized, Placebo Controlled, Dose Escalating, Parallel Group Study To Investigate The Safety, Toleration And Pharmacokinetics Of Single Doses Of PF-04418948 In Healthy Male Subjects
Brief Title: A Study To Investigate The Safety And Toleration Of A Single Dose Of PF-04418948 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B0631001
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
MeSH Terms: interventions — 1-(4-fluorobenzoyl)-3-(((6-methoxy-2-naphthyl)oxy)methyl)azetidine-3-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- PF-04418948 30 mg (Experimental)
  Interventions: Drug: PF-04418948
- PF-04418948 100 mg (Experimental)
  Interventions: Drug: PF-04418948
- PF-04418948 300 mg (Experimental)
  Interventions: Drug: PF-04418948
- PF-04418948 1000 mg (Experimental)
  Interventions: Drug: PF-04418948
- PF-04418948 3000 mg (Experimental)
  Interventions: Drug: PF-04418948
- PF-04418948 4500 mg (Experimental)
  Interventions: Drug: PF-04418948
- PF-04418948 6000 mg (Experimental)
  Interventions: Drug: PF-04418948

INTERVENTIONS:
Drug: PF-04418948 — solution, 30 mg, single
  Arms: PF-04418948 30 mg
Drug: PF-04418948 — solution, 100 mg, single
  Arms: PF-04418948 100 mg
Drug: PF-04418948 — solution, 300 mg, single
  Arms: PF-04418948 300 mg
Drug: PF-04418948 — solution, 1000 mg, single
  Arms: PF-04418948 1000 mg
Drug: PF-04418948 — solution, 3000 mg, single
  Arms: PF-04418948 3000 mg
Drug: PF-04418948 — solution, 4500 mg, single
  Arms: PF-04418948 4500 mg
Drug: PF-04418948 — solution, 6000 mg, single
  Arms: PF-04418948 6000 mg

SUMMARY:
The purpose of this study is to investigate safety and toleration of single oral doses as well as the time course of PF-04418948 concentration in the blood following dosing by oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week for males.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters: Cmax, Tmax, AUClast, AUCtau, AUCinf, Cav, CL/F, V/F, t1/2 | 240 hours
Safety: Adverse events, vital signs measurements, telemetry, 12-lead ECGs, physical examination findings, blood safety tests, fecal occult blood (FOB), cardiac troponin measurements, urine safety tests (KIM-1 measurements and creatinine). | 240 hours

SECONDARY OUTCOMES:
Pharmacodynamics: Emax (maximum observed increase in TNFα concentration from pre-dose level) TEmax (time to Emax), AUEClast, AUECt (where t will be a defined timepoint) and maximum n-fold increase in concentration from pre-dose level. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0631001&StudyName=A%20Study%20To%20Investigate%20The%20Safety%20And%20Toleration%20Of%20A%20Single%20Dose%20Of%20PF-04418948%20In%20Healthy%20Volunteers